CLINICAL TRIAL: NCT00253760
Title: Metabolic Analysis in Human Sulfur Amino Acid Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R03 DK66008 (completed 2007); R03DK066008 (NIH)
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Oxidative Stress; Diabetes; Heart Diseases
Keywords: redox; sulfur amino acids; glutathione; aging
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases | interventions — Cysteine; Methionine

INTERVENTIONS:
Drug: dietary amino acids; cysteine and methionine

SUMMARY:
Varied food intake, disease, and genetic differences result in complex diet-health interactions. In principle, information-rich metabolic analyses combined with bioinformatic tools provide an approach to explore these interactions. This project is a feasibility study of the use of high-resolution 1H-nuclear magnetic resonance (NMR) to study metabolic perturbations induced by a deficiency in sulfur amino acids (SAA). The investigators will 1) test the hypothesis that deficient dietary intake of SAA in humans results in oxidation of reduced glutathione (GSH)/oxidized glutathione (GSSG) redox and 2) determine whether 1H-NMR of blood and urine detects metabolic changes due to SAA deficiency.

DETAILED DESCRIPTION:
Varied food intake, disease, and genetic differences result in complex diet-health interactions. In principle, information-rich metabolic analyses combined with bioinformatic tools provide an approach to explore these interactions. This project is a feasibility study of the use of high-resolution 1H-NMR to study metabolic perturbations induced by deficiency in sulfur amino acids (SAA). In cell culture, sulfur amino acid (SAA) deficiency results in substantial oxidation of glutathione (GSH) redox state. Because GSH redox affects central homeostatic and cell defense mechanisms, redox changes in vivo due to SAA deficiency could induce complex physiologic effects that are not easily predictable by more traditional metabolic analyses. We will 1) test the hypothesis that deficient dietary intake of SAA in humans results in oxidation of GSH/GSSG redox and 2) determine whether 1H-NMR of blood and urine detects metabolic changes due to SAA deficiency. Studies will be performed on 12 healthy individuals (6 males, 6 females) in the Emory General Clinical Research Center (GCRC) using a crossover design (replete, deficient, replete). Kinetic and balance studies will establish the time course and magnitude of changes in SAA and metabolites in blood and urine in response to SAA intake. Plasma GSH/GSSG and cysteine/cystine redox will be measured to determine whether variation in intake of SAA affects steady-state thiol-disulfide redox state. 1H-NMR spectra of blood and urine samples will be used to determine whether metabolic changes unrelated to the direct SAA metabolites can be detected in association with variation in SAA intake. The results will show whether variation in SAA intake is likely to affect health risks associated with thiol-disulfide redox and oxidative stress. Furthermore, because NMR analysis of biofluids can be performed with a high throughput (e.g., 300 samples/day with a flow cell), results will show whether this approach could be useful for nutritional assessment of complex metabolic effects of SAA intake.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight
* Males or females

Exclusion Criteria:

* Smokers
* Pregnancy
* Chronic illness other than hypertension
* Age less than 18 and greater than 40 years

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2004-02; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
redox state of the two central low molecular weight thiol-disulfide pools, i.e., GSH/GSSG and cysteine (Cys)/cystine (CySS)
a global metabolic spectrum detectable by H-NMR

CONTACTS AND LOCATIONS:
Overall Officials: Dean P Jones, Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States